CLINICAL TRIAL: NCT03270696
Title: Efficacy of Neuromuscular Blockade Before Facemask Ventilation in Inducing General Anesthesia
Brief Title: Simultaneous Injection of Propofol and Rocuronium in Inducing General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Hwa Seo, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JHSeo_MV
Record Dates: First submitted 2017-08-23; First posted 2017-09-01 (Actual); Last update posted 2018-04-12 (Actual); Status verified 2017-09

CONDITIONS: Anesthesia; Functional
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- simultaneous administration of propofol and rocuronium (Experimental): In this group, the investigator will administrate propofol (2ml/kg) and rocuronium (0.6mg/kg) simultaneously, and start facemask ventilation after patient loss consciousness to induce general anesthesia.
  The investigator will measure the mean tidal volume (TV) applied during facemask ventilation for 1 minute.
  Interventions: Drug: administration of propofol and rocuronium
- ordinal administration of propofol and rocuronium (Experimental): In this group, the investigator will administrate propofol (2ml/kg) first, and follow injection of rocuronium (0.6mg/kg) after patient loss consciousness and confirming facemask ventilation.
  The investigator will measure the mean tidal volume (TV) applied during facemask ventilation for 1 minute.
  Interventions: Drug: administration of propofol and rocuronium

INTERVENTIONS:
Drug: administration of propofol and rocuronium — compare the tidal volume applied from starting facemask ventilation under 15cmH2O of PCV for 1 minute according to administrating propofol and rocuronium simultaneously, or ordinally

SUMMARY:
This study is conducted to evaluate the efficacy of simultaneous injection of propofol and rocuronium in inducing general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective surgery requiring endotracheal intubation
* ASA I, II, and III
* above 20 years

Exclusion Criteria:

* refuse to enroll
* patients with risk of aspirating gastric contents
* patients in whom NMBs are contraindicated
* patients with predictors of difficult mask ventilation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
mean tidal volume | from starting facemask ventilation for 1 minute
  mean tidal volume of facemask ventilation in 1 minute

CONTACTS AND LOCATIONS:
Overall Officials: JH Seo, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Min SH, Im H, Kim BR, Yoon S, Bahk JH, Seo JH. Randomized Trial Comparing Early and Late Administration of Rocuronium Before and After Checking Mask Ventilation in Patients With Normal Airways. Anesth Analg. 2019 Aug;129(2):380-386. doi: 10.1213/ANE.0000000000004060. PMID 30768462